CLINICAL TRIAL: NCT02686411
Title: A Prospective Evaluation of Satisfaction With Quality of Care on the Palliative Care Unit
Brief Title: Evaluation of Satisfaction With Quality of Care on the Palliative Care Unit
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1074; NCI-2020-11433 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-1074 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-02-17; First posted 2016-02-19 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey): Patients and caregivers complete surveys over 5-10 minutes before and after care in the PCU.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study examines the difference between the quality of care patients receive with palliative care consult services and the palliative care unit. This may help researchers learn how improvements can be made to the level of care provided in the palliative care unit and improve satisfaction with quality of care by patients and caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the change of satisfaction with quality of care after an experience on the palliative care unit (PCU) for both patients and caregivers, as determined by the global rating survey.

SECONDARY OBJECTIVES:

I. To determine the change of the quality of care as determined by patients and caregivers utilizing validated assessment tools and a global rating survey assessing different aspects of care after PCU.

II. To determine domains of care that are strongly or poorly provided by the PCU, as reported by patient and caregiver opinions on quality of care.

III. To determine which demographic features (i.e. cancer diagnosis; time since diagnosis; reason for transfer to the PCU; gender; caregiver ethnic group; comfort with the idea of transfer to the PCU; Memorial Delirium Assessment Scale [MDAS], Edmonton Symptom Assessment Scale [ESAS], and distress thermometer) may correlate with patient and caregiver satisfaction with PCU care measured by global survey and with the family satisfaction with end-of-life care.

OUTLINE:

Patients and caregivers complete surveys over 5-10 minutes before and after care in the PCU.

ELIGIBILITY:
Inclusion Criteria:

* Patients and/or patients' caregivers who have completed at least 2 weekdays on an in-patient service together with the assistance of the palliative care consult services (PCCS), and who then are transitioned to the care of the PCU team along with an admission order to that effect
* A caregiver (if participating) must have been present with the patient during 2 weekdays on the inpatient service and present for at least 2 weekdays of care on the PCU
* Both patient and caregiver participation is optional but both must be 18 years of age or older
* A caregiver will be defined by the patient as "the person most involved with their care". However, if the patient lacks capacity, the caregiver will be decided via discussion with individuals indicated in the patient's Medical Power of Attorney or the Texas rule of law if this is not present
* Both patient and caregiver (if participating) must understand, read and speak English
* Both patient (if actively participating) and caregiver (if participating) must sign an informed consent form

Exclusion Criteria:

* Patients or caregivers with physical limitations (visual or motor impairment) causing inability to read, complete or sign the consent form and surveys after considering appropriate aid and assistance
* Patients or caregivers who the research staff, bedside nurse, or palliative care physician or mid-level provider deems unable to participate due to poor cognitive capacity or acute physical distress
* Caregivers who are not able to attend the patient for at least 2 weekdays while on the PCU
* Patients who are imminently dying as determined by the palliative physician (or designated advanced practice provider [APP]/fellow)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and/or patients' caregivers who have completed at least 2 weekdays on an in-patient service together
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Relative satisfaction rate | through study completion, an average of 1 year
  Defined as the percentage of patients that answered "Better" and "Much Better" to the first question in the global rating on "overall care". The relative satisfaction rate after palliative care unit (PCU) care in patients or caregivers will be estimated with 95% confidence interval.
Patient Global Survey/Caregiver Global Survey | through study completion, an average of 1 year
  Assessed by Edmonton Symptom Assessment Scale (ESAS), Memorial Delirium Assessment Scale (MDAS) distress thermometer will be summarized by descriptive analysis and/or tabulation.
Distress thermometer | through study completion, an average of 1 year
  Measured by Family Satisfaction with end-of-life care will be summarized descriptively for each time point and may be compared within patients and within caregivers before and after the PCU by Wilcoxon signed-rank test, when the outcome is on Likert ordinal scales with 3, 5 levels or even 10 levels and the differences in the scales can be considered as continuous variables.
Patients' and caregivers' opinions on quality of care | through study completion, an average of 1 year
  Measured by Family Satisfaction with end-of-life care will be summarized descriptively for each time point and may be compared within patients and within caregivers before and after the PCU by Wilcoxon signed-rank test, when the outcome is on Likert ordinal scales with 3, 5 levels or even 10 levels and the differences in the scales can be considered as continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan Azhar, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org